CLINICAL TRIAL: NCT01086150
Title: Use of Topical Lidocaine (Lidoderm 5% Patch) to Reduce Pain in Patients With Diabetic Neuropathy: Does the Density and Subtype of Sodium Channels Affect Response?
Brief Title: Use of Topical Lidocaine to Reduce Pain in Patients With Diabetic Neuropathy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Albany Medical College (Other)
Collaborators: Endo Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Charles Argoff, MD, Albany Medical College
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENDO
Record Dates: First submitted 2010-03-11; First posted 2010-03-12 (Estimated); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Diabetic Peripheral Neuropathy
MeSH Terms: interventions — Lidocaine; Transdermal Patch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy control patients (Other): Subjects 18 to 70 years of age, non-diabetic with no nervous system disease. Lidocaine 5% patch applied to both feet daily, Skin biopsies at biaseline and end of study.
  Interventions: Procedure: Skin biopsy; Drug: Lidocaine 5% patches
- Type I or Type II diabetes with painful diabetic neuropathy (Other): 18 to 70 years old with significantly painful diabetic neuropathy.Lidocaine 5% patch applied to both feet daily, Skin biopsies at biaseline and end of study.
  Interventions: Procedure: Skin biopsy; Drug: Lidocaine 5% patches
- patients with non-painful diabetic peripheral neuropathy (Other): 18-70 years of age with Type I or Type II diabetes with non-painful or insignificantly painful diabetic neuropathy.Lidocaine 5% patch applied to both feet daily, Skin biopsies at baseline, 4 weeks, and end of study.
  Interventions: Procedure: Skin biopsy; Drug: Lidocaine 5% patches

INTERVENTIONS:
Procedure: Skin biopsy — Skin biopsy specimens will processed and analyzed for Nerve fiber count, nerve and skin morphology, and sodium channel specific epitope expression in keratinocytes.
Drug: Lidocaine 5% patches — Subject will apply patches to affected area QD for 12 hours then remove.

SUMMARY:
The purpose of this study is to see if an investigational drug known as the lidocaine 5% patch is safe and effective in reducing the symptoms of diabetic neuropathy, to examine how topical lidocaine affects the nerve endings, and to determine whether treatment with the lidocaine patch can prevent the potential progression to chronic diabetic neuropathy pain in subjects who did not report pain at the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: 18-70 years of age, non-diabetic with no nervous system disease (healthy control group)
* Group 2: 18-70 years of age with Type I or Type II diabetes with significantly painful diabetic neuropathy (VAS > 40mm at Baseline)
* Group 3: 18-70 years of age with Type I or Type II diabetes with non- painful or insignificantly painful diabetic neuropathy (VAS < 40mm at Baseline)

Exclusion Criteria:

* History of clinically significant liver disease, serious peripheral vascular disease, a blood clotting disorder, or any other medical condition felt to be exclusionary by the investigator
* Allergy to lidocaine
* Unwillingness to sign informed consent or any other reasons for which the investigator feels the subject cannot complete the study
* Women who are pregnant, breastfeeding or trying to become pregnant
* History of slow-healing diabetic foot ulcers
* Current skin or soft tissue lesions on the foot that will interfere with application of the lidocaine patch and or skin biopsies
* Subjects taking Class I antiarrhythmics
* HgA1c > 11%
* Active cancer within the previous two years except treated basal cell carcinoma of the skin
* Co-morbidities that can produce neuropathy
* Subjects taking sodium channel blockers within one week of study treatment and throughout the study
* Subjects taking any other experimental drugs within 30 days prior to Screening Visit (Visit 1)
* Application of lidocaine patch to either foot within two weeks of Screening Visit (Visit 1)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Albany Medical College, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Control Patients | Type I or Type II Diabetes With Painful Diabetic Neuropathy | Patients With Non-painful Diabetic Peripheral Neuropathy
Started | 11 | 27 | 13
Completed | 11 | 21 | 12
Not Completed | 0 | 6 | 1
Not completed — Withdrawal by Subject | 0 | 4 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Screen Failure | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Control Patients | Type I or Type II Diabetes With Painful Diabetic Neuropathy | Patients With Non-painful Diabetic Peripheral Neuropathy | Total
Number analyzed (Participants) | 11 | 21 | 12 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 19 | 10 | 40
  >=65 years | 0 | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 4 | 19
  Male | 5 | 12 | 8 | 25

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores From Composite Visual Analog Scale
Description: Scores range from 0 to 10 with higher scores indicating higher levels of pain.
Time Frame: baseline, 4 weeks
Population: Healthy controls were not assessed for this measure.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Healthy Control Patients | Type I or Type II Diabetes With Painful Diabetic Neuropathy | Patients With Non-painful Diabetic Peripheral Neuropathy
Number analyzed (Participants) | 0 | 21 | 12
units on a scale
  Baseline |  | 6.5 [4.5 to 9] | 1.2 [0 to 3.1]
  4 weeks |  | 4.5 [0 to 8.9] | 0.5 [0 to 1.5]

2. Secondary Outcome: Keratinocyte Immunoreactivity of Nav1.6, Nav1.7, CGRP
Description: Pixel intensity (0-256) of immunofluorescence for each individual biomarker.
Time Frame: Baseline, 4 weeks
Measure: Mean (Full Range); unit: Pixel intensity (0-256)
Arm/Group | Healthy Control Patients | Type I or Type II Diabetes With Painful Diabetic Neuropathy | Patients With Non-painful Diabetic Peripheral Neuropathy
Number analyzed (Participants) | 11 | 21 | 12
Pixel intensity (0-256)
  Nav1.6-baseline | 81.2 [63.54 to 127.38] | 101.4 [64.69 to 135.5] | 87.9 [49.3 to 126.44]
  Nav1.6-4 weeks | 91 [49.19 to 132.37] | 90.7 [60.85 to 134.63] | 90.8 [60.38 to 148.07]
  Nav1.7-baseline | 47.5 [30.84 to 73.33] | 59.6 [39.41 to 87.53] | 54.3 [40.66 to 66.9]
  Nav1.7-4 weeks | 52.4 [39.82 to 85.83] | 51.5 [30.3 to 81.35] | 54.7 [34.43 to 77.57]
  CGRP-baseline | 27.7 [22.37 to 32.83] | 38.5 [27.49 to 68.14] | 29.5 [19.51 to 39.83]
  CGRP-4 weeks | 31.5 [21.86 to 49.53] | 32.8 [19.03 to 56.1] | 26.2 [20.52 to 36.58]

ADVERSE EVENTS:
Arm/Group | Healthy Control Patients | Type I or Type II Diabetes With Painful Diabetic Neuropathy | Patients With Non-painful Diabetic Peripheral Neuropathy
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/21 | 0/12
Other Adverse Events (participants affected / at risk) | 0/11 | 0/21 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No